CLINICAL TRIAL: NCT01075815
Title: Exploratory Study to Determine the Effect of Lutropin Alfa on Embryo Quality and Their Implantation in Women of Advanced Reproductive Age
Brief Title: A Clinical Trial to Determine the Effect of Lutropin Alfa on Embryo Quality and Implantation Rate in Advanced Reproductive Age
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 700642-500; 2008-002281-55 (EudraCT Number)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Infertility; Ovulation Induction
Keywords: Infertility; Ovulation induction; Luveris; Controlled ovarian stimulation; Reproductive technologies, assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFSH + rhLH (Experimental): Recombinant human luteinizing hormone (rhLH,Luveris®) injection 150 IU subcutaneously daily along with rFSH 300 IU subcutaneously daily from S1 to S4 and then rFSH dose can be adjusted depending on the ovarian response till r-hCG administration day.
  Interventions: Drug: Recombinant human luteinizing hormone (rhLH); Drug: Recombinant follicle-stimulating hormone (rFSH)
- rFSH (Active Comparator): rFSH injection 300 IU subcutaneously daily from S1 to S4 and then dose can be adjusted depending on the ovarian response till r-hCG administration day.
  Interventions: Drug: Recombinant follicle-stimulating hormone (rFSH)

INTERVENTIONS:
Drug: Recombinant human luteinizing hormone (rhLH)
  Other Names: Luveris®; Lutropin alfa
  Arms: rFSH + rhLH
Drug: Recombinant follicle-stimulating hormone (rFSH)

SUMMARY:
This is a multicentric, open, randomized, comparative trial aimed to assess the influence of recombinant luteinizing hormone (r-LH) supplementation during controlled ovarian stimulation (COS) in advanced reproductive age in terms of improved embryo competence which allows to transfer less embryos to avoid high grade multiple pregnancy without reducing the pregnancy rate.

DETAILED DESCRIPTION:
This study will be carried out by the Grupo de Interés de Salud Embrionaria (GISE) group (part of the Spanish Fertility Society) who uses strict criteria to select the embryos most suitable for successful transference.

OBJECTIVES

Primary objective:

* To determine the benefit of r-LH supplementation in COS prior to in-vitro fertilization (IVF)/intracytosolic sperm injection (ICSI) in advanced reproductive age, in terms of embryo competence to implant, as compared against no r-LH supplementation

Secondary objectives:

To evaluate the benefit of r-LH supplementation in COS, in terms of:

* follicular development
* length of the stimulation
* oocyte number and their maturity
* fertilization rate
* embryo number and quality
* gestational sacs
* abortion
* ongoing pregnancies
* local and systemic safety of r-LH administration

The study will consist of 2 groups randomized in 1:1 ratio and each subject would be followed up until the confirmation of her pregnancy status. Each subject will be administered gonadotropin releasing hormone (GnRH) agonist subcutaneously daily from previous mid luteal phase to r-hCG administration as a standard practice to achieve down regulation. Each subject will also be administered recombinant follicle stimulating hormone (r-FSH) at a starting dose of 300 IU from S1 up to ovarian stimulation completion (r-hCG day) as a part of standard practice. In addition to the above concurrent therapies, one group will be administered experimental treatment (Luveris®) and the other group (control group) will not be administered any other drug (control treatment) during the stimulation period from stimulation start (S1) up to ovarian stimulation completion or stimulation cancellation respectively. Ovarian stimulation on an average takes 11 days and it is expected that stimulation period will not be extended beyond 15 days. A single injection of r-hCG will be administered intramuscularly or subcutaneously after the last injection of Luveris or r-FSH to achieve final follicular maturation. After, 34-36 hours of administration of r-hCG OPU will be done for oocyte retrieval and embryo transfer (ET) will be conducted within 5 days from OPU. Subjects will also be provided luteal support with natural progesterone and will be followed until delivery or miscarriage. Ultrasound and estradiol (E2) assessment of follicular growth will be conducted at various time points during the stimulation period with or without treatment adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female subject aged greater than (>) 35 years
* Subjects with baseline FSH serum level less than or equal to (<=) 10 IU/liter (l), LH and E2 levels within local normal range and plasma prolactin levels < 30 nanogram/milliliter (ng/ml)
* Subjects with regular spontaneous menstrual cycles of 25-35 days
* Subjects with infertility justifying IVF/ICSI-ET treatment
* Subjects programmed for COS with r-FSH under GnRH agonist protocol
* Sperm from current male partner suitable for IVF/ICSI according to local lab, unless sperm donor is foreseen
* Subjects with presence of both ovaries
* Subjects whose uterine cavity is able to sustain embryo implantation or pregnancy
* Subjects with normal papanicolaou test (PAP) smear within previous 3 years
* Subjects with body mass index (BMI) < 30 at stimulation start
* Subjects who receive confirmation of not being pregnant by a negative beta-hCG test (urine or blood) prior to starting r-FSH administration
* Subjects willing and able to comply with the protocol for the duration of the study
* Subjects who have given informed consent prior to any study-related procedure not part of normal medical care

Exclusion Criteria:

* Subjects or her male partners who are known to be human immunodeficiency virus, hepatitis B virus or hepatitis C virus positive
* Subjects with any clinically significant systemic disease; tumors of the hypothalamus and pituitary gland; ovarian, uterine or mammary cancer; hormonal abnormality and/or medical, biochemical, hematological condition which in the judgment of the investigator may interfere with gonadotropin treatment
* Subjects with more than 2 previous assisted reproductive technologies (ART) cycles
* Subjects in which previous cycles were cancelled due to poor response (< 3 antral follicles after 15 day of stimulation)
* Subjects with cryopreserved embryos from previous ART cycles
* Subjects with unexplained gynecological bleeding
* Subjects with polycystic ovaries, ovarian enlargement or cyst of unknown etiology
* Subjects known to have any contraindication to being pregnant and/or carrying pregnancy to term
* Subjects with known allergy to gonadotrophin preparations or any of the excipients
* Subjects known to have any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years
* Subjects with previous entry into this study or simultaneous participation in another clinical drug trial
* Subjects who have refused to or inability to comply with the protocol

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck, S.L., Spain
Locations (1):
- FivMadrid, C/ Marqués de Urquijo, 26,, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One out of 76 randomized participants did not receive study medication.
Groups:
- rFSH + rhLH: Recombinant human luteinizing hormone (rhLH, Luveris®) injection 150 International Units (IU) subcutaneously daily along with recombinant follicle-stimulating hormone (rFSH) 300 IU subcutaneously daily from Day 1 of stimulation period (S1) to Day 4 of stimulation period (S4) and then rFSH dose adjusted depending on the ovarian response till recombinant human choriogonadotropin (r-hCG) administration day.
- rFSH: Recombinant follicle stimulating hormone (rFSH) injection 300 IU subcutaneously daily from S1 to S4 and then dose adjusted depending on the ovarian response till r-hCG administration day.
Period: Overall Study
Arm/Group | rFSH + rhLH | rFSH
Started | 40 (Number of participants treated.) | 35 (Number of participants treated.)
Completed | 30 | 31
Not Completed | 10 | 4
Not completed — Withdrawal before r-hCG administration | 6 | 1
Not completed — Withdrawal between rhCG-ovum pickup(OPU) | 1 | 1
Not completed — Withdrawal between OPU - embryo transfer | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFSH + rhLH | rFSH | Total
Number analyzed (Participants) | 40 | 35 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (2.2) | 37.3 (1.5) | 37.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Implantation Rate
Description: Implantation rate was measured as the number of gestational sacs observed, divided by the number of embryos transferred.
Time Frame: Day 35-42 post ovum pick-up (OPU) (34-38 hours post recombinant human choriogonadotropin day {end of stimulation cycle}[approximately 28 days])
Population: Intention to treat (ITT) population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: sacs per embryo
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
sacs per embryo | 0.2 (0.4) | 0.2 (0.3)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.8762, Wilcoxon two sample test; Mean Difference (Final Values) = 0.0235, 95% CI 2-sided [-0.1546 to 0.1568]

2. Secondary Outcome: Mean Number of Follicles Greater Than or Equal to 14 Millimeter (mm) on Recombinant Human Choriogonadotropin (r-hCG) Day
Time Frame: r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
follicles | 7.7 (4.9) | 8.7 (4.0)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.3589, ANOVA

3. Secondary Outcome: Mean Number of Oocytes Retrieved
Description: Mean number of oocytes retrieved per reporting group on the day of OPU (34-38 hours post r-hCG day (end of stimulation cycle [approximately 28 days]) was calculated. Oocyte retrieval is a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Time Frame: 34-38 hours post r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
oocytes | 5.9 (3.9) | 7.7 (4.0)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.0629, Wilcoxon two sample test

4. Secondary Outcome: Number of Mature Oocytes Retrieved
Description: Number of mature oocytes retrieved per reporting group on the day of OPU (34-38 hours post r-hCG day (end of stimulation cycle [approximately 28 days]) was calculated. Oocyte retrieval is a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body. The nuclear maturity was evaluated based on the presence of a germinal vesicle (GV) or whether oocytes were in metaphase I (Meta-I) or II (Meta-II) stage.
Time Frame: 34-38 hours post r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: mature oocytes
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
mature oocytes | 234 | 271
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.4728, ANOVA

5. Secondary Outcome: Number of Fertilized Oocytes (2 Pronuclei [PN])
Description: Oocytes were fertilized using Intra-cytoplasmic Sperm Injection (ICSI) technique which is an in-vitro fertilization procedure in which a single sperm is injected directly into an egg under a microscope. The appearance of two 2PN is the first sign of successful fertilization as observed during in vitro fertilization, and is usually observed after ICSI. The zygote is then termed 2PN.
Time Frame: 34-38 hours post r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: 2PN oocytes
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
2PN oocytes | 128 | 136
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.0950, Fisher Exact

6. Secondary Outcome: Number and Quality of Embryos
Description: Embryos were graded according to Spanish Association for the Study of Reproductive Biology (ASEBIR) criteria into different categories: (A) optimal quality with maximum capacity for implantation, (B) good quality with a high capacity for implantation, (C) regular with low possibility of implantation and (D) poor quality with very little possibility of implantation.
Time Frame: Day 2-3 post OPU (34-38 hours post r-hCG day {end of stimulation cycle}[approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication. Here "N" represents the number of participants who had at least one fertilized oocyte.
Measure: Number; unit: embyros
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 31 | 32
embyros
  A + B (good quality) | 69 | 65
  C + D (poor quality) | 56 | 73
  Total embryos | 125 | 138

7. Secondary Outcome: Number of Participants With Biochemical Pregnancies
Description: Biochemical pregnancy was defined as a pregnancy diagnosed only by the detection of hCG in serum or urine and that does not develop into a clinical pregnancy.
Time Frame: 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
participants | 11 | 10
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.9179, Chi-squared; Risk Ratio (RR) = 0.9625, 95% CI 2-sided [0.4655 to 1.9900]

8. Secondary Outcome: Number of Participants With Clinical Pregnancies
Description: Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.
Time Frame: 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
participants | 10 | 10
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.7271, Chi-squared; Risk Ratio (RR) = 0.8750, 95% CI 2-sided [0.4133 to 1.8524]

9. Secondary Outcome: Total Dose of Recombinant Follicle Stimulating Hormone (r-FSH)
Time Frame: 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
IU | 2812.2 (719.4) | 2970.3 (748.2)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.3267, Wilcoxon two sample test

10. Secondary Outcome: Estradiol (E2) Levels on r-hCG Day
Time Frame: r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication. Here "N" represents the number of participants with plasma E2 levels at r-hCG day.
Measure: Mean (Standard Deviation); unit: picogram/milliter (pg/mL)
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 33 | 29
picogram/milliter (pg/mL) | 1890.2 (1084.4) | 1621 (827.8)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.4164, Wilcoxon two sample test

11. Secondary Outcome: Number of Ovarian Stimulation Days
Description: Ovarian stimulation included from first rFSH injection (S1) until day on which r-hCG was administered (r-hCG day). This period was divided into 2 parts: the first period in which 300 International Unit (IU) rFSH dose was constant and which covered from S1 to Day 4 of stimulation period (S4); the second period in which the rFSH dose could be adjusted depending on the ovarian response and which began on S4 and finished on the day on which the criteria for administration of r-hCG to induce the final follicular maturation were met.
Time Frame: S1 up to r-hCG day (end of stimulation cycle [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
Days | 9.7 (2.1) | 9.8 (1.9)
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.5952, Wilcoxon two sample test

12. Secondary Outcome: Number of Recombinant Human Choriogonadotropin (r-hCG) Cycles Cancelled Due to Poor Response
Description: Poor response was defined as 3 or less follicles of greater than or equal to 12 mm developing following at least 7 days of study treatment.
Time Frame: Up to 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication.
Measure: Number; unit: cycles
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
cycles | 4 | 1

13. Secondary Outcome: Total Number of Births
Description: Total number of births per reporting group was calculated.
Time Frame: Up to 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: ITT population included all randomized participants who had received at least 1 dose of the study medication. Here "N" represents number of participants evaluated for this measure.
Measure: Number; unit: births
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 34
births | 10 | 9
Statistical Analysis 1: Comparison: rFSH + rhLH vs rFSH; Test type: Superiority or Other; p = 0.8852, Chi-squared; Risk Ratio (RR) = 0.9444, 95% CI 2-sided [0.4347 to 2.0518]

14. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: Safety population included all participants who had received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
participants | 19 | 9

15. Secondary Outcome: Number of Participants With Ovarian Hyper Stimulation Syndrome (OHSS)
Description: OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, hemoconcentration, and increased blood clotting.
Time Frame: Baseline up to 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: Safety population included all participants who had received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
participants | 1 | 0

16. Secondary Outcome: Number of Cycles Cancelled Due to Risk of Ovarian Hyper Stimulation Syndrome (OHSS)
Description: as for outcome 15
Time Frame: Baseline up to 2 months after OPU (34-38 hours post r-hCG day {end of stimulation cycle} [approximately 28 days])
Population: Safety population included all participants who had received at least 1 dose of the study medication.
Measure: Number; unit: cycles
Arm/Group | rFSH + rhLH | rFSH
Number analyzed (Participants) | 40 | 35
cycles | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs are collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until the post-treatment safety, on day 35-42 post-hCG administration. AEs are classified as pre-treatment, treatment-emergent and post-treatment.
Description: Pre-Treatment:Medical conditions present at the initial study visit that did not worsen in severity or frequency during the study;Treatment-Emergent: If the onset date of the AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of the AE was post-hCG Days 35- 42 for participants who completed the study.
Arm/Group | rFSH + rhLH | rFSH
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/35
Other Adverse Events (participants affected / at risk) | 17/40 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFSH + rhLH (N=40) | rFSH (N=35)
New born hip dysplasia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cutaneous anginoma (Skin and subcutaneous tissue disorders) | 1 | 0
Trisomy 13 (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFSH + rhLH (N=40) | rFSH (N=35)
Premature birth (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 1 | 2
Bloating (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 1 | 2
Pain at the injection site (General disorders) | 5 | 0
Erythema at the injection site (General disorders) | 2 | 0
Pruritus at the injection site (General disorders) | 2 | 0
Haematoma (Vascular disorders) | 4 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Genital secretion (Reproductive system and breast disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Haematoma at the injection site (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 1
Inflammation at the injection site (General disorders) | 1 | 0
General malaise (General disorders) | 1 | 0
Reaction at the injection site (General disorders) | 1 | 0
Mood change (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other